CLINICAL TRIAL: NCT03317886
Title: Mesenteric Approach vs. Conventional Approach for Pancreatic Cancer During Pancreaticoduodenectomy (MAPLE-PD Trial)
Brief Title: Mesenteric Approach vs. Conventional Approach for Pancreatic Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Hiroki Yamaue, Professor, Wakayama Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2128
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreaticoduodenectomy; Mesenteric Approach
MeSH Terms: interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mesenteric approach (Active Comparator): mesenteric approach starts from lymph node dissection around the superior mesenteric artery and performs Kocher's maneuver finally during pancreaticoduodenectomy.
  Interventions: Procedure: pancreaticoduodenectomy
- conventional approach (Active Comparator): Conventional approach starts from Kocher's maneuver and finally performs lymph node dissection around the superior mesenteric artery during pancreaticoduodenectomy.
  Interventions: Procedure: pancreaticoduodenectomy

INTERVENTIONS:
Procedure: pancreaticoduodenectomy — pancreaticoduodenectomy for pancreatic ductal adenocarcinoma

SUMMARY:
The aim of this study is to evaluate the advantage of mesenteric approach during pancreaticoduodenectomy (PD) for pancreatic ductal adenocarcinoma (PDAC). The design of this study is multicenter randomized clinical trial, comparing oncological and surgical outcomes between mesenteric approach and conventional approach during PD for PDAC.

DETAILED DESCRIPTION:
Mesenteric approach starts from dissection of lymph nodes around the superior mesenteric artery (SMA) and finally performs Kocher's maneuver during PD. The aims of this approach are 1) decrease of intraoperative blood loss volume, 2) increase of R0 rate, and 3) prevention of squeezing cancer cells out into the vessels. However, there have been no evidence of the efficacy of this procedure. Therefore, the aim of this study is to evaluate the efficacy of mesenteric approach during PD for PDAC, by multicenter randomized clinical trial comparing oncological and surgical outcomes between mesenteric approach and conventional approach during PD for PDAC.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who are scheduled to undergo pancreaticoduodenectomy for resectable or borderline resectable (only portal vein invasion) pancreatic ductal adenocarcinoma.
2. Patients whose Eastern Cooperative Oncology Group performance status are 0 or 1.
3. Patients who are 20 years or older.
4. Patients who have adequate organ function.
5. Patients who understand sufficiently the study to provide written informed consent

Exclusion Criteria:

1. Patients who have severe ischemic cardiovascular disease
2. Patients who have liver cirrhosis or active hepatitis
3. Patients who need oxygen due to interstitial pneumonia or lung fibrosis
4. Patients who receive dialysis due to chronic renal failure
5. Patients who need surrounding organ resection
6. Patients who need artery reconstruction
7. Patients who are diagnosed as positive para-aortic lymph node metastases based on preoperative imaging
8. Patients who have active multiple cancer that is thought to influence the occurrence of adverse events
9. Patients who take steroid for the long period that is thought to influence the occurrence of adverse events
10. Patients who undergo laparoscopic or laparoscopy-assisted pancreaticoduodenectomy
11. Patients who cannot understand ths study due to psychotic disease or psychological symptoms
12. Patients whose preoperative biopsy tissues are diagnosed as other pathological findings than pancreatic ductal adenocarcinoma
13. Patients who underwent gastrectomy or colon/ rectum resection previously
14. Patients who have severe drug allergy to iodine and gadolinium

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | up to 48 months
  survival from surgery to death

SECONDARY OUTCOMES:
operative time | up to 24 months
  time for operation
time for resection | up to 3 months
  time for resection
intraoperative blood loss | up to 3 months
  intraoperative blood loss volume
blood transfusion volume | up to 3 months
  transfusion volume required during operation
grade B/C pancreatic fistula rate | up to 3 months
  grade B/C pancreatic fistula rate according to International Study Group of Pancreatic Surgery (ISGPS) definition
rate of delayed gastric emptying | up to 3 months
  rate of delayed gastric emptying according to International Study Group of Pancreatic Surgery (ISGPS) definition
abdominal hemorrhage rate | up to 3 months
  abdominal hemorrhage rate according to International Study Group of Pancreatic Surgery (ISGPS) definition
all morbidity rate | up to 3 months
  rate of all postoperative complications
mortality rate | up to 3 months
  rate of operative death
diarrhea rate | up to 24 months
  rate of postoperative rate
R0 rate | up to 3 months
  pathological R0 rate
R1 rate | up to 3 months
  pathological R1 rate
the closest length between surgical margin and cancer cell | up to 3 months
  the closest length between surgical margin and cancer cell if R0
number of harvested lymph nodes | up to 3 months
  number of harvested lymph nodes
number of metastatic lymph nodes | up to 3 months
  number of metastatic lymph nodes
lymph node ratio | up to 3 months
  number of metastatic lymph nodes divided by number of harvested lymph nodes
recurrence free survival | up to 24 months
  survival from operation date to recurrence date
site of initial recurrence | up to 24 months
  site of initial recurrence

CONTACTS AND LOCATIONS:
Locations (15):
- Japan (15):
  - Kyusyu University, Fukuoka
  - Kansai Medical University, Hirakata
  - Hiroshima University, Hiroshima
  - Shimane University, Izumo
  - Kagoshima University, Kagoshima
  - Nara Medical University, Kashihara
  - Kumamoto University, Kumamoto
  - Nagoya University, Nagoya
  - Osaka Medical University, Osaka
  - Osaka University, Osaka
  - Shiga Medical University, Ōtsu
  - Kinki University, Sayama
  - Tokyo Medical University, Tokyo
  - Toyama University, Toyama
  - Wakayama Medical University, Wakayama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hirono S, Kitahata Y, Motobayashi H, Satoi S, Sho M, Takami H, Kamei K, Shibuya K, Hidaka M, Uemura K, Kimura K, Mataki Y, Nagakawa Y, Hayashi H, Morimura R, Nakamura M, Wan K, Shimokawa T, Nakao A, Yamaue H; MAPLE-PD trial investigators. Mesenteric Versus Conventional Approach During Pancreatoduodenectomy for Pancreatic Ductal Adenocarcinoma (MAPLE-PD trial): A Multicenter Randomized Controlled Trial. Ann Surg. 2025 Aug 7. doi: 10.1097/SLA.0000000000006900. Online ahead of print. PMID 40772617
- [Derived] Hirono S, Kawai M, Okada KI, Fujii T, Sho M, Satoi S, Amano R, Eguchi H, Mataki Y, Nakamura M, Matsumoto I, Baba H, Tani M, Kawabata Y, Nagakawa Y, Yamada S, Murakami Y, Shimokawa T, Yamaue H. MAPLE-PD trial (Mesenteric Approach vs. Conventional Approach for Pancreatic Cancer during Pancreaticoduodenectomy): study protocol for a multicenter randomized controlled trial of 354 patients with pancreatic ductal adenocarcinoma. Trials. 2018 Nov 8;19(1):613. doi: 10.1186/s13063-018-3002-z. PMID 30409152